CLINICAL TRIAL: NCT03268577
Title: Interactive Diet and Activity Tracking in AARP (IDATA): Biomarker Based Validation Study of Internet-Based and Conventional Self-Report Instruments for Assessing Diet and Physical Activity Within AARP
Brief Title: Internet-Based and Self-Reports in Assessing Diet and Physical Activity Within AARP
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2017-01184; NCI-2017-01184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11CN155 (Other: NCI Division of Cancer Control and Population Sciences); DCP-003 (Other: DCP)
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, urine, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prevention (diet and activity tracking): Patients complete the ASA24 about foods, cooking methods, and other aspects of diet every 2 months for up to 6 times, and complete ACT24 about activities and time reporting every 2 months for up to 6 times. Patients also complete DHQ-II questionnaires at the beginning and end of the study about the frequency and portion sizes of foods consumed over the past 12 months, provide a 7-day food checklist twice with the DHQ-II, and provide a 4-day food record twice, once every 6 months. Physical activity monitors are worn to measure movement at different intensity levels and sitting or standing periods, twice during the study with 6 months between each time they are worn.
  Interventions: Other: Internet-Based Intervention; Device: Monitoring Device; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Complete ASA24
Other: Internet-Based Intervention — Complete ACT24 reporting
Device: Monitoring Device — Wear accelerometer and inclinometer physical activity monitors
  Other Names: Monitor
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies how well internet-based and self-report instruments measure food intake and physical activity levels and their relationship with disease within American Association of Retired Persons (AARP) members. Comparing new internet-based questionnaires developed by the National Cancer Institute that report all the foods consumed and activities performed in an entire day to standardized physical measurements may help to determine if the information collected is accurate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the measurement error structure of self-reported dietary assessment instruments, including, a food frequency questionnaire (National Cancer Institute [NCI]'s Diet History Questionnaire-II [DHQ-II]), and 24-hour recalls using the new automated self-administered 24-hour dietary recall (ASA24) instrument with respect to absolute energy intake, absolute protein intake, and protein density-and potentially other nutritional factors such as potassium intake.

II. Investigate the measurement error structure associated with self-reported active and sedentary behaviors, including multiple administrations of a new 24-hour recall (activity completed over time in 24-hours [ACT24]) and selected questionnaires using energy expenditure from doubly labeled water (DLW) and physical activities measures of physical activity monitors as reference instruments.

III. Evaluate alternative analytic approaches for combining different types of self-report data on diet and physical activity-related behaviors as well as self-report plus objective data (derived from activity monitors, heart rate monitors e.g.).

IV. Within the context of an AARP-based cohort, explore the adjustment of observed RRs for several key cancer hypotheses related to diet and physical activity based on the measurement error data provided by the new study.

V. Evaluate the potential for 'energy adjustment' that incorporates physical activity and body size.

OUTLINE:

Patients complete the ASA24 about foods, cooking methods, and other aspects of diet every 2 months for up to 6 times, and complete ACT24 about activities and time reporting every 2 months for up to 6 times. Patients also complete DHQ-II questionnaires at the beginning and end of the study about the frequency and portion sizes of foods consumed over the past 12 months, provide a 7-day food checklist twice with the DHQ-II, and provide a 4-day food record twice, once every 6 months. Physical activity monitors are worn to measure movement at different intensity levels and sitting or standing periods, twice during the study with 6 months between each time they are worn.

ELIGIBILITY:
Exclusion Criteria:

* Non-English speaking or reading
* Weight loss diet (liquid or medications)
* Diabetes
* Body mass index < 18.5 or >= 40 (kg/m^2)
* History of renal failure, congestive heart failure, or other conditions involving disturbances in fluid balance
* Limited mobility
* Use of supplemental oxygen
* Allergy to para-amino benzoic acid (PABA)
* No access to high-speed internet
* No more than one AARP member in the household can participate in the study

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members within the existing NIH-AARP Diet and Health Study members (aged 50-71 in 1995-96) and younger AARP members born after 1945 ('baby boomers') and living in the Pittsburgh area in Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Self-reported energy intake from automated self-administered 24-hour dietary recall (ASA24), Diet History Questionnaire (DHQ)-II, and 4-day food record | Up to 12 months
  Will be evaluated against energy intake measured by doubly labeled water (DLW). Dietary intake of protein, potassium, and other nutrients will be compared to urinary nitrogen (UN), urinary potassium, and other nutrients measured in urine and blood.
Measurement error structure of self-reported active and sedentary behaviors (e.g. activity completed over time in 24-hours [ACT24], questionnaires) | Up to 12 months
  Will be examined using energy expenditure measured by DLW, physical activity monitor data, and hear rate monitor data. Data will be also used to evaluate alternative statistical methods for combining different types of self-report data on diet and physical activity-related behaviors as well as self-report plus objectively measured data.
24-hour urine samples | Up to 12 months
  Will be analyzed for UN, potassium, para-amino benzoic acid (PABA), and other nutrients that are potential objective markers of intakes. First morning void urine also will be evaluated for its potential to be used as a source of biomarkers replacing 24-hr urine. Urine will be analyzed to characterize metabolic profiles of individuals.
Fasting blood sample analyses | Up to 12 months
  Will be processed to extract plasma and red and white blood cells, and analyzed in the future for vitamin C, folate, vitamin E, vitamin A, carotenoids, lipids, fatty acids and other nutrients.
Saliva samples | Up to 12 months
  Will be analyzed for oral microbiomes and to characterize metabolic profiles of individuals.
Measurement error structure of self-reported dietary assessment instruments | Up to 12 months
  Evaluated using latent-variable (measurement error) models. The models allow self-reported dietary intake to have intake-related and person-specific biases, but assume that reference biomarkers (doubly-labeled water, urinary nitrogen, urinary potassium) provide unbiased estimates of true usual intake at the individual level. Such models allow one to estimate the joint distribution of true and reported intake, and to estimate parameters of interest such as the correlation of true and reported intake and the "attenuation factor", or slope in the regression of true intake on reported intake.
Measurement error in self-reported total physical activity (measured in energy expenditure) | Up to 12 months
  Evaluated using latent-variable (measurement error) models. The models allow total energy expenditure derived from a physical activity monitor to have intake-related and person-specific biases, but assume that reference biomarkers (doubly-labeled water, urinary nitrogen, urinary potassium) provide unbiased estimates of true usual intake at the individual level. Such models to help develop better algorithms for estimating total energy expenditure from the measurements of physical activity monitors. For other physical activity measures of interest, such as minutes of vigorous activity or minutes of sedentary time per day, will use the physical activity monitors to derive approximately unbiased estimates that can be used as reference instruments.
Reduction in measurement error | Up to 12 months
  Will use multivariate measurement error models to estimate the joint distribution of true and reported values (nutrient intake, total energy, physical activity, body size). Then calculate residual reported intake (given reported total energy, physical activity and body size) and residual true intake (given true total energy, physical activity and body size), and assess the measurement error properties of reported residual intake as a measure of true residual intake. Specifically, will calculate the correlation of true and reported residual intake and the attenuation factor for residual reported intake and compare them to the same measures calculated for the simpler model that adjusts only for energy.

CONTACTS AND LOCATIONS:
Overall Officials: heather bowles, Principal Investigator — NCI Division of Cancer Control and Population Sciences
Locations (1):
- NCI Division of Cancer Control and Population Sciences, Rockville, Maryland, United States

REFERENCES:
- [Derived] Chang DC, Dodd KW, Abramowitz MK, Barrett B, Stinson EJ. Validation of Net Endogenous Acid Production from the Automated Self-Administered 24-h Recall, 4-d Food Records, and a Food Frequency Questionnaire Using Urine Markers. J Nutr. 2025 Jun 30:S0022-3166(25)00402-X. doi: 10.1016/j.tjnut.2025.06.017. Online ahead of print. PMID 40602721
- [Derived] Abar L, Steele EM, Lee SK, Kahle L, Moore SC, Watts E, O'Connell CP, Matthews CE, Herrick KA, Hall KD, O'Connor LE, Freedman ND, Sinha R, Hong HG, Loftfield E. Identification and validation of poly-metabolite scores for diets high in ultra-processed food: An observational study and post-hoc randomized controlled crossover-feeding trial. PLoS Med. 2025 May 20;22(5):e1004560. doi: 10.1371/journal.pmed.1004560. eCollection 2025 May. PMID 40392756
- [Derived] Chang DC, Stinson EJ, Dodd KW, Bowles HR, Herrick KA, Schoeller DA, Barrett B, Votruba SB, Krakoff J, Kavouras SA. Validation of Total Water Intake from the Automated Self-Administered 24-h Recall, 4-d Food Records, and a Food Frequency Questionnaire Using Doubly Labeled Water. J Nutr. 2023 Oct;153(10):3049-3057. doi: 10.1016/j.tjnut.2023.08.027. Epub 2023 Sep 3. PMID 37660952
- [Derived] Shams-White MM, Korycinski RW, Dodd KW, Barrett B, Jacobs S, Subar AF, Park Y, Bowles HR. Examining the association between meal context and diet quality: an observational study of meal context in older adults. Int J Behav Nutr Phys Act. 2021 May 20;18(1):67. doi: 10.1186/s12966-021-01122-x. PMID 34016140
- [Derived] Subar AF, Potischman N, Dodd KW, Thompson FE, Baer DJ, Schoeller DA, Midthune D, Kipnis V, Kirkpatrick SI, Mittl B, Zimmerman TP, Douglass D, Bowles HR, Park Y. Performance and Feasibility of Recalls Completed Using the Automated Self-Administered 24-Hour Dietary Assessment Tool in Relation to Other Self-Report Tools and Biomarkers in the Interactive Diet and Activity Tracking in AARP (IDATA) Study. J Acad Nutr Diet. 2020 Nov;120(11):1805-1820. doi: 10.1016/j.jand.2020.06.015. Epub 2020 Aug 17. PMID 32819883